CLINICAL TRIAL: NCT06244550
Title: A Clinical Trial Using Ganwei (HepatoKeeper) Herbal Essentials to Treat Non-Alcoholic Fatty Liver Disease
Brief Title: Clinical Trials Using HepatoKeeper Herbal Essentials to Treat Non-alcoholic Fatty Liver Disease and Metabolic Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Collaborators: The One Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: TCHIRB-11002006
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Non-alcoholic Fatty Liver Disease; Liver Fibrosis; Liver Injury
Keywords: Ganwei; Non-alcoholic fatty liver disease; metformin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo + metformin (Experimental): Double blinded: matching placebo + metformin
  Placebo daily metformin 1500mg daily
  Interventions: Drug: Metformin; Drug: Placebo
- Ganwei + metformin (Experimental): Double blinded: Ganwei + metformin
  Ganwei 500mg/15 kg of body weight, daily metformin 1500mg daily
  Interventions: Drug: Ganwei; Drug: Metformin
- Placebo (Placebo Comparator): Double blinded: matching placebo
  Placebo daily
  Interventions: Drug: Placebo
- Ganwei (Experimental): Double blinded: Ganwei
  Ganwei 500mg/15 kg of body weight, daily
  Interventions: Drug: Ganwei

INTERVENTIONS:
Drug: Ganwei — Capsules
  Other Names: HepatoKeeper
  Arms: Ganwei; Ganwei + metformin
Drug: Metformin — Tablets
  Other Names: A10BA02
  Arms: Ganwei + metformin; Placebo + metformin
Drug: Placebo — Matching capsules
  Arms: Placebo; Placebo + metformin

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common liver disease globally, with an estimated prevalence of approximately 15 to 30%. The incidence of NAFLD is even higher, reaching up to 58%, in individuals who are overweight or obese. The pathogenesis of NAFLD is complex and not fully understood. The metabolism of carbohydrates contributes to the development of NAFLD, as it increases the enzymatic activity of lipid synthesis in the liver, depleting adenosine triphosphate (ATP) rapidly and causing stress on mitochondria and endoplasmic reticulum. The multifunctional protein Glycine N-methyltransferase (GNMT) plays a regulatory role in liver carbohydrate metabolism, and its expression is downregulated in the liver tissues of NAFLD.

While weight loss and lifestyle adjustments are helpful in controlling NAFLD, effective pharmacological or healthcare interventions for NAFLD patients are currently lacking. Insulin resistance is crucial in the pathogenesis of NAFLD, suggesting that drugs improving insulin sensitivity, such as metformin, might have therapeutic effects. However, recent large-scale clinical trial results have not supported this hypothesis. Investigators propose that the mitochondrial inhibitory effects of metformin may be related to this discrepancy, and the negative effects may be reversed through food containing substances promoting GNMT gene expression, such as Ganwei (as know as "HepatoKeeper"). Preliminary animal experiments also show that the combined use of metformin and GNMT enhancers effectively eliminates liver lipid droplet accumulation and improves liver inflammation in a NAFLD mouse model, surpassing the effects of either drug used alone.

Based on these findings, our team designed the medication treatment group for this clinical trial, aiming to investigate whether the combination of Ganwei and metformin produces a synergistic effect in humans. Ganwei compound herbal extract capsules contain extracts from natural foods such as Schisandra chinensis, Paeonia lactiflora, and Punica granatum. Among them, Paeonia lactiflora is known to contain components that enhance GNMT expression. Animal and cell experiments have demonstrated its potential for repairing liver damage and inflammation. This trial aims to assess the impact of orally administering Ganwei compound herbal extract capsules on participants and evaluate its effects on fatty liver, liver fibrosis, and metabolic indicators.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common liver disease globally, with an estimated prevalence of approximately 15 to 30%. The incidence of NAFLD is even higher, reaching up to 58%, in individuals who are overweight or obese (Schwenger, 2014). With the Westernization of diets and insufficient physical activity, the prevalence of obesity, diabetes, and hyperlipidemia has been increasing in Taiwan in recent years, contributing to the gradual rise in the prevalence of NAFLD. NAFLD is strongly associated with metabolic syndrome, cardiovascular diseases, insulin resistance, and may progress to hepatitis, liver fibrosis, and even cirrhosis (Fazel, 2016; Amr, 2020).

The pathogenesis of NAFLD is complex and not fully understood. Current understanding suggests that environmental factors such as diet, exercise, obesity, gut microbiota, and genetics play a role in the development of NAFLD. The liver, responsible for metabolizing major substances including carbohydrates and fatty acids, becomes overwhelmed, leading to the production of toxic lipids. Disruptions in lipid metabolism, inhibition of mitochondrial function, and impaired export of triglycerides from liver cells contribute to the accumulation of lipids within the liver. Insulin resistance further exacerbates this process. Additionally, lipid alterations in liver cells increase oxidative stress and activate cell signaling, triggering immune responses that damage liver cells and contribute to the development of fatty liver inflammation, fibrosis, and potentially liver cancer (Fazel, 2016; Amr, 2020).

The metabolism of carbohydrates also contributes to NAFLD, as it increases the enzymatic activity of lipid synthesis in the liver, depleting adenosine triphosphate (ATP) rapidly and causing stress on mitochondria and endoplasmic reticulum. This results in liver cell necrosis, contributing to the development of NAFLD. The multifunctional protein Glycine N-methyltransferase (GNMT) plays a regulatory role in liver carbohydrate metabolism, and its expression is downregulated in the liver tissues of NAFLD (Liao, 2012).

While weight loss and lifestyle adjustments are helpful in controlling NAFLD, effective pharmacological or healthcare interventions for NAFLD patients are currently lacking (Julien et al., 2019; Mary et al., 2020). Insulin resistance is crucial in the pathogenesis of NAFLD, suggesting that drugs improving insulin sensitivity, such as metformin, might have therapeutic effects. However, recent large-scale clinical trial results have not supported this hypothesis. Investigators propose that the mitochondrial inhibitory effects of metformin may be related to this discrepancy, and the negative effects may be reversed through food containing substances promoting GNMT gene expression, such as Ganwei (as know as "HepatoKeeper"). Preliminary animal experiments also show that the combined use of metformin and GNMT enhancers effectively eliminates liver lipid droplet accumulation and improves liver inflammation in a NAFLD mouse model, surpassing the effects of either drug used alone.

Based on these findings, our team designed the medication treatment group for this clinical trial, aiming to investigate whether the combination of Ganwei and metformin produces a synergistic effect in humans. Ganwei compound herbal extract capsules contain extracts from natural foods such as Schisandra chinensis, Paeonia lactiflora, and Punica granatum. Among them, Paeonia lactiflora is known to contain components that enhance GNMT expression (Kyu-Han et al., 2020; Rajni et al., 2019). Animal and cell experiments have demonstrated its potential for repairing liver damage and inflammation. This trial aims to assess the impact of orally administering Ganwei compound herbal extract capsules on participants and evaluate its effects on fatty liver, liver fibrosis, and metabolic indicators.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to participate in the study and provide written informed consent.
* Male and female adults ≥20 and <80 years of age.
* Suspected or confirmed diagnosis of NAFLD:

  * Fibroscan with CAP ≥220 dB/m
  * Criteria for diagnosing fatty liver: Abdominal ultrasound reveals differences in liver and kidney parenchyma due to wave reflection, liver parenchymal ultrasound attenuation, and blurred imaging of liver vessels and diaphragm, indicating fatty liver.

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding.
* Diabetic patients undergoing medication treatment.
* Patients clinically diagnosed with alcoholic hepatitis, autoimmune hepatitis, or biliary liver disease.
* Excessive alcohol consumption (more than 15 grams/day for females, more than 30 grams/day for males).
* Users of weight-loss products and vitamin E supplements.
* Individuals with an estimated Glomerular Filtration Rate (eGFR) less than 60 mL/min/1.73m².

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Liver steatosis severity: the change of CAP (dB/m) by Fibroscan | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Controlled Attenuation Parameter(CAP) by FibroScan
Liver fibrosis severity: the change of kPa by Fibroscan | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in kPa by FibroScan

SECONDARY OUTCOMES:
Aspartate Transaminase (AST) | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Aspartate Transaminase (AST)
Alanine amino Transferase (ALT) | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Alanine amino Transferase (ALT)
Body mass index (BMI) | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Body mass index (BMI)
Glycated Hemoglobin (HbA1c) | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Glycated Hemoglobin (HbA1c)
White blood cell (WBC) | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in White blood cell (WBC)
C-reactive protein (CRP) | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in C-reactive protein (CRP)
Triglyceride (TG) | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Triglyceride (TG)
estimated Glomerular filtration rate (eGFR) | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in estimated Glomerular filtration rate (eGFR)
Physical functioning | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Physical functioning by 36-Item Short Form Health Survey (SF-36)
Role limitations due to physical health | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Role limitations due to physical health by 36-Item Short Form Health Survey (SF-36)
Role limitations due to emotional problems | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Role limitations due to emotional problems by 36-Item Short Form Health Survey (SF-36)
Energy/fatigue | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Energy/fatigue by 36-Item Short Form Health Survey (SF-36)
Emotional well-being | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Emotional well-being by 36-Item Short Form Health Survey (SF-36)
Social functioning | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Social functioning by 36-Item Short Form Health Survey (SF-36)
Bodily pain | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in Pain by 36-Item Short Form Health Survey (SF-36)
General health | Week 24
  The effect of once daily, oral administration of 500 mg/15 kg of body weight Ganwei and/or 1500 mg metformin 24 weeks treatment versus before on the change in General health by 36-Item Short Form Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Lin Lin, MD., Principal Investigator — Department of Gastroenterology, Renai branch, Taipei City Hospital, Taipei, Taiwan.
Locations (1):
- Taipei City Hospital, Taipei, Taiwan